CLINICAL TRIAL: NCT05723445
Title: The Effects of a Low Glycemic Load Diet on Dysglycemia and Body Composition in Adults With Cystic Fibrosis-Related Diabetes
Acronym: DINE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1943156-3
Record Dates: First submitted 2023-01-16; First posted 2023-02-10 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Cystic Fibrosis; Cystic Fibrosis-related Diabetes; Cystic Fibrosis With Intestinal Manifestations
Keywords: Cystic Fibrosis-Related Diabetes; Low Glycemic Load; Continuous Glucose Monitoring; Body Composition
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: Single dietary treatment with a meal-delivery phase and free-living conditions phase, as well as a run-in period as a control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Low Glycemic Load Diet (Experimental): Feeding study with dietary composition (approximately) 50% fat, 20% protein, 30% carbohydrate.
  Interventions: Behavioral: Low Glycemic Load Diet

INTERVENTIONS:
Behavioral: Low Glycemic Load Diet — Food delivery service will provide a low glycemic load diet for 8 weeks, followed by a 4-month period of self-adherence to a low glycemic load diet with close nutritionist follow up

SUMMARY:
This study will evalute the effect of a low glycemic load (LGL diet on dysglycemia, insulin requirements, DXA-derived body composition, gastrointestinal symptoms and quality of life measures in adults with cystic fibrosis-related diabetes (CFRD). We will use continuous glucose monitors (CGM) to assess the LGL diet both in a controlled setting (via a meal delivery company) and in free-living conditions.

DETAILED DESCRIPTION:
Maintenance of a healthy body mass index (BMI) is a well-established marker of improved morbidity and mortality in patients with cystic fibrosis (CF). To achieve and maintain adequate weight, patients with CF are encouraged to consume a caloric intake of 120-150% of the dietary reference intake (DRI) for the typical healthy adult. However, dietary recommendations for children and adults with CF are based entirely on consensus and expert opinion. High carbohydrate intake is typical for patients with CF, but this may lead to multiple complications including post-prandial hyperglycemia, increased inflammation, and abnormal GI motility and may predispose to obesity and metabolic syndrome. Dietary changes are a commonly used treatment approach for CF-related diabetes (CFRD), despite the fact that there are no data establishing whether dietary interventions are helpful in preventing and/or treating CFRD. Particularly as patients with CF live longer with highly effective modulator therapy and as the prevalence of cardiovascular and metabolic disease increases in this population, it is crucial to understand the effects of dietary composition on short and long-term endocrine, GI, and pulmonary outcomes.

In patients with both type 1 and type 2 diabetes mellitus, a low glycemic load (LGL) diet has been shown to improve glycemic variability, A1c level, insulin sensitivity, and quality of life without increasing hypoglycemic events. Significant glycemic variability is associated with increased markers of inflammation in adolescents with T1DM, possibly serving as a mechanistic link to the development of cardiovascular disease. Particularly as rates of obesity and cardiovascular disease continue to increase, this diet may be particularly useful in patients with CF, altered glucose homeostasis, and/or obesity. There are currently no prospective studies evaluating the impact of diet quality on glycemic control and body composition in patients with CF. The gold standard approach for assessing the safety and efficacy of dietary interventions is a food delivery study.

The investigators will conduct a prospective, open-label study in adults with CFRD to determine the effects of an LGL diet on dysglycemia and body composition. Participants will initially follow their standard diet for a 10-day run-in period. They will then transition to an LGL diet provided by a meal delivery company for 8 weeks. During this period, they will wear a continuous glucose monitor (CGM) for 2 10-day periods. Finally, participants will adhere to an LGL diet under free-living conditions with close nutritionist follow-up for a period of 4 months. Serum studies, DXA-body composition, anthropometric data, GI symptoms and quality of life measures will be obtained at baseline, after the meal-delivery phase and at study completion.

The investigators hypothesize that an LGL diet will result in improved CGM-derived measures of hyperglycemia, a decrease in insulin requirements, and reductions in fat-mass index on DXA analysis in adults with CFRD over an 8-week period during a meal delivery period. Furthermore, they hypothesize that these changes will be sustainable under free-living conditions during a 4-month period.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and above
* Genetically confirmed diagnosis of CF
* Diagnosis of pancreatic insufficiency, requiring pancreatic enzyme replacement
* Criteria for CFRD:

A.) Most recent OGTT 2-hour glucose >200 mg/dL within the past two years, and/or; B.) HbA1c >6.5% in the past two years, and/or; C.) Current use of insulin

Exclusion Criteria:

* FEV1 <50% predicted on most recent pulmonary function testing
* BMI <18 kg/m2
* Currently receiving enteral nutrition support via GT feeds
* Pregnancy, plan to become pregnant in the next 3-months, or sexually active without use of contraception
* Use of IV antibiotics or systemic supraphysiologic glucocorticoids for CF exacerbation within 1 month
* Started or stopped treatment with a CFTR modulator within 3 months of enrollment
* Currently adhering to an LGL or other carbohydrate-restricted diet (carbohydrate intake <30% of total daily caloric intake)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in percent time in target range 70-180 mg/dL | Baseline, post-meal delivery phase (8 weeks), post-free-living conditions phase (4 months)
  Continuous glucose monitoring

SECONDARY OUTCOMES:
Change in CGM average glucose (AG) mg/dL | Baseline, post-meal delivery phase (8 weeks), post-free-living conditions phase (4 months)
  Continuous glucose monitoring
Change in percent time >180 mg/dL | Baseline, post-meal delivery phase (8 weeks), post-free-living conditions phase (4 months)
  Continuous glucose monitoring
Change in percent time >250 mg/dL | Baseline, post-meal delivery phase (8 weeks), post-free-living conditions phase (4 months)
  Continuous glucose monitoring
Change in CGM standard deviation (SD) | Baseline, post-meal delivery phase (8 weeks), post-free-living conditions phase (4 months)
  Continuous glucose monitoring
Change in CGM coefficient of variation (CV) | Baseline, post-meal delivery phase (8 weeks), post-free-living conditions phase (4 months)
  Continuous glucose monitoring
Change in percent time <70 mg/dL | Baseline, post-meal delivery phase (8 weeks), post-free-living conditions phase (4 months)
  Continuous glucose monitoring
Change in percent time <54 mg/dL | Baseline, post-meal delivery phase (8 weeks), post-free-living conditions phase (4 months)
  Continuous glucose monitoring
Change in number of episodes of symptomatic hypoglycemia (average per week) | Baseline (weeks 1-2), visit 2 (post-meal delivery phase, weeks 2-10), visit 3 (post-free living conditions phase, weeks 11-26))
  Weekly emailed survey
Change in total daily dose of insulin (TDD) | Baseline (weeks 1-2), visit 2 (post-meal delivery phase, weeks 2-10), visit 3 (post-free living conditions phase, weeks 11-26)
  Weekly emailed survey
Change in body mass index (BMI, kg/m2) | Baseline (weeks 1-2), visit 2 (post-meal delivery phase, weeks 2-10), visit 3 (post-free living conditions phase, weeks 11-26)
  Every other week emailed survey
Change in weight (kg) | Baseline (weeks 1-2), visit 2 (post-meal delivery phase, weeks 2-10), visit 3 (post-free living conditions phase, weeks 11-26)
  Every other week emailed survey
Change fat-mass index (FMI, fat mass kg/ height m^2) | Baseline (week 1), visit 2 (post-meal delivery phase, week10), visit 3 (post-free living conditions phase, week 26)
  DXA body composition measures
Change in percent body fat (%) | Baseline (week 1), visit 2 (post-meal delivery phase, week10), visit 3 (post-free living conditions phase, week 26)
  DXA body composition measures
Change in appendicular lean mass index (ALMI, lean mass kg/ height m^2) | Baseline (week 1), visit 2 (post-meal delivery phase, week10), visit 3 (post-free living conditions phase, week 26)
  DXA body composition measures
Change in Patient Assessment of Constipation (PAC) questionnaire score | Baseline (week 1), visit 2 (post-meal delivery phase, week10), visit 3 (post-free living conditions phase, week 26)
  Likert scale questionnaire with 12 items, each scored 0-4, total score ranging from 0-48 with higher scores related to worse outcomes
Change in Patient Assessment of Gastrointestinal Symptoms (PAGI-Sym) questionnaire score | Baseline (week 1), visit 2 (post-meal delivery phase, week10), visit 3 (post-free living conditions phase, week 26)
  Likert scale questionnaire with 20 items, each scored 0-5, total score ranging from 0-100 with higher scores related to worse outcomes
Change in Cystic Fibrosis Questionnaire Revised (CFQ-R) score | Baseline (week 1), visit 2 (post-meal delivery phase, week10), visit 3 (post-free living conditions phase, week 26)
  Likert scale questionnaire with 50 items, each scored 0-4, total score ranging from 0-100 with higher scores reflecting better outcomes
Change in Diet Tolerability Questionnaire | Baseline (week 1), visit 2 (post-meal delivery phase, week10), visit 3 (post-free living conditions phase, week 26)
  Likert scale questionnaire with 5 items, each scored 0-10, total score ranging from 0-50 with higher scores reflecting better diet tolerability
Change in Bristol stool chart data | Baseline (week 1), visit 2 (post-meal delivery phase, week10), visit 3 (post-free living conditions phase, week 26)
  Chart depicting 7 types of stool patterns, ranging from constipation to diarrhea
Change in erythrocyte sedimentation rate (ESR) | Baseline (week 1), visit 2 (post-meal delivery phase, week10), visit 3 (post-free living conditions phase, week 26)
  Laboratory test, measured in mm/hr
Change in c-reactive protein (CRP) | Baseline (week 1), visit 2 (post-meal delivery phase, week10), visit 3 (post-free living conditions phase, week 26)
  Laboratory test, measured in mg/L
Change in hemoglobin A1c | Baseline (week 1), visit 2 (post-meal delivery phase, week10), visit 3 (post-free living conditions phase, week 26)
  Laboratory test, measured in %
Change in total cholesterol | Baseline (week 1), visit 2 (post-meal delivery phase, week10), visit 3 (post-free living conditions phase, week 26)
  Laboratory test, measured in mg/dL
Change in high-density lipoprotein (HDL) | Baseline (week 1), visit 2 (post-meal delivery phase, week10), visit 3 (post-free living conditions phase, week 26)
  Laboratory test, measured in mg/dL
Change in low-density lipoprotein (LDL) | Baseline (week 1), visit 2 (post-meal delivery phase, week10), visit 3 (post-free living conditions phase, week 26)
  Laboratory test, measured in mg/dL
Change in triglyceride level | Baseline (week 1), visit 2 (post-meal delivery phase, week10), visit 3 (post-free living conditions phase, week 26)
  Laboratory test, measured in mg/dL
Change in intestinal fatty acid binding protein (I-FABP) | Baseline (week 1), visit 2 (post-meal delivery phase, week10), visit 3 (post-free living conditions phase, week 26)
  Laboratory test, measured in ng/mL

CONTACTS AND LOCATIONS:
Overall Officials: Kevin J Scully, MB BCh BAO, Principal Investigator — Rhode Island Hospital; Melissa S Putman, MD, MSc, Principal Investigator — Boston Children's Hospital
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Rhode Island Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD data with other researchers

REFERENCES:
- [Background] Culhane S, George C, Pearo B, Spoede E. Malnutrition in cystic fibrosis: a review. Nutr Clin Pract. 2013 Dec;28(6):676-83. doi: 10.1177/0884533613507086. Epub 2013 Oct 29. PMID 24170579
- [Background] Moran A, Brunzell C, Cohen RC, Katz M, Marshall BC, Onady G, Robinson KA, Sabadosa KA, Stecenko A, Slovis B; CFRD Guidelines Committee. Clinical care guidelines for cystic fibrosis-related diabetes: a position statement of the American Diabetes Association and a clinical practice guideline of the Cystic Fibrosis Foundation, endorsed by the Pediatric Endocrine Society. Diabetes Care. 2010 Dec;33(12):2697-708. doi: 10.2337/dc10-1768. No abstract available. PMID 21115772
- [Background] Gaskin KJ. Nutritional care in children with cystic fibrosis: are our patients becoming better? Eur J Clin Nutr. 2013 May;67(5):558-64. doi: 10.1038/ejcn.2013.20. Epub 2013 Mar 6. PMID 23462946
- [Background] Thomas D, Elliott EJ. Low glycaemic index, or low glycaemic load, diets for diabetes mellitus. Cochrane Database Syst Rev. 2009 Jan 21;2009(1):CD006296. doi: 10.1002/14651858.CD006296.pub2. PMID 19160276
- [Background] Hoffman RP, Dye AS, Huang H, Bauer JA. Glycemic variability predicts inflammation in adolescents with type 1 diabetes. J Pediatr Endocrinol Metab. 2016 Oct 1;29(10):1129-1133. doi: 10.1515/jpem-2016-0139. PMID 27658133
- [Background] Panagopoulou P, Fotoulaki M, Nikolaou A, Nousia-Arvanitakis S. Prevalence of malnutrition and obesity among cystic fibrosis patients. Pediatr Int. 2014 Feb;56(1):89-94. doi: 10.1111/ped.12214. PMID 24003895
- [Background] Stephenson AL, Mannik LA, Walsh S, Brotherwood M, Robert R, Darling PB, Nisenbaum R, Moerman J, Stanojevic S. Longitudinal trends in nutritional status and the relation between lung function and BMI in cystic fibrosis: a population-based cohort study. Am J Clin Nutr. 2013 Apr;97(4):872-7. doi: 10.3945/ajcn.112.051409. Epub 2013 Feb 6. PMID 23388659
- [Background] Harindhanavudhi T, Wang Q, Dunitz J, Moran A, Moheet A. Prevalence and factors associated with overweight and obesity in adults with cystic fibrosis: A single-center analysis. J Cyst Fibros. 2020 Jan;19(1):139-145. doi: 10.1016/j.jcf.2019.10.004. Epub 2019 Nov 11. PMID 31727452
- [Background] Lennerz BS, Barton A, Bernstein RK, Dikeman RD, Diulus C, Hallberg S, Rhodes ET, Ebbeling CB, Westman EC, Yancy WS Jr, Ludwig DS. Management of Type 1 Diabetes With a Very Low-Carbohydrate Diet. Pediatrics. 2018 Jun;141(6):e20173349. doi: 10.1542/peds.2017-3349. Epub 2018 May 7. PMID 29735574
- [Background] Norris AW, Ode KL, Merjaneh L, Sanda S, Yi Y, Sun X, Engelhardt JF, Hull RL. Survival in a bad neighborhood: pancreatic islets in cystic fibrosis. J Endocrinol. 2019 Apr;241(1):R35-R50. doi: 10.1530/JOE-18-0468. PMID 30759072
- [Background] Prentice BJ, Ooi CY, Strachan RE, Hameed S, Ebrahimkhani S, Waters SA, Verge CF, Widger J. Early glucose abnormalities are associated with pulmonary inflammation in young children with cystic fibrosis. J Cyst Fibros. 2019 Nov;18(6):869-873. doi: 10.1016/j.jcf.2019.03.010. Epub 2019 Apr 26. PMID 31036487
- [Background] Ode KL, Frohnert B, Laguna T, Phillips J, Holme B, Regelmann W, Thomas W, Moran A. Oral glucose tolerance testing in children with cystic fibrosis. Pediatr Diabetes. 2010 Nov;11(7):487-92. doi: 10.1111/j.1399-5448.2009.00632.x. PMID 20202149
- [Background] Bellissimo MP, Zhang I, Ivie EA, Tran PH, Tangpricha V, Hunt WR, Stecenko AA, Ziegler TR, Alvarez JA. Visceral adipose tissue is associated with poor diet quality and higher fasting glucose in adults with cystic fibrosis. J Cyst Fibros. 2019 May;18(3):430-435. doi: 10.1016/j.jcf.2019.01.002. Epub 2019 Jan 18. PMID 30665857
- [Background] Scully KJ, Sherwood JS, Martin K, Ruazol M, Marchetti P, Larkin M, Zheng H, Sawicki GS, Uluer A, Neuringer I, Yonker LM, Sicilian L, Wexler DJ, Putman MS. Continuous Glucose Monitoring and HbA1c in Cystic Fibrosis: Clinical Correlations and Implications for CFRD Diagnosis. J Clin Endocrinol Metab. 2022 Mar 24;107(4):e1444-e1454. doi: 10.1210/clinem/dgab857. PMID 34850006
- [Background] Scully KJ, Jay LT, Freedman S, Sawicki GS, Uluer A, Finkelstein JS, Putman MS. The Relationship between Body Composition, Dietary Intake, Physical Activity, and Pulmonary Status in Adolescents and Adults with Cystic Fibrosis. Nutrients. 2022 Jan 12;14(2):310. doi: 10.3390/nu14020310. PMID 35057491
- [Background] Sheikh S, Zemel BS, Stallings VA, Rubenstein RC, Kelly A. Body composition and pulmonary function in cystic fibrosis. Front Pediatr. 2014 Apr 15;2:33. doi: 10.3389/fped.2014.00033. eCollection 2014. PMID 24783186
- [Background] Vargas S, Romance R, Petro JL, Bonilla DA, Galancho I, Espinar S, Kreider RB, Benitez-Porres J. Efficacy of ketogenic diet on body composition during resistance training in trained men: a randomized controlled trial. J Int Soc Sports Nutr. 2018 Jul 9;15(1):31. doi: 10.1186/s12970-018-0236-9. PMID 29986720
- [Background] Gorji Z, Modaresi M, Yekanni-Nejad S, Mahmoudi M. Effects of low glycemic index/high-fat, high-calorie diet on glycemic control and lipid profiles of children and adolescence with cystic fibrosis: A randomized double-blind controlled clinical trial. Diabetes Metab Syndr. 2020 Mar-Apr;14(2):87-92. doi: 10.1016/j.dsx.2019.12.010. Epub 2020 Jan 8. PMID 31991298
- [Background] Riddlesworth TD, Beck RW, Gal RL, Connor CG, Bergenstal RM, Lee S, Willi SM. Optimal Sampling Duration for Continuous Glucose Monitoring to Determine Long-Term Glycemic Control. Diabetes Technol Ther. 2018 Apr;20(4):314-316. doi: 10.1089/dia.2017.0455. Epub 2018 Mar 22. PMID 29565197
- [Background] Scully KJ, Marchetti P, Sawicki GS, Uluer A, Cernadas M, Cagnina RE, Kennedy JC, Putman MS. The effect of elexacaftor/tezacaftor/ivacaftor (ETI) on glycemia in adults with cystic fibrosis. J Cyst Fibros. 2022 Mar;21(2):258-263. doi: 10.1016/j.jcf.2021.09.001. Epub 2021 Sep 14. PMID 34531155
- [Background] Marquis P, De La Loge C, Dubois D, McDermott A, Chassany O. Development and validation of the Patient Assessment of Constipation Quality of Life questionnaire. Scand J Gastroenterol. 2005 May;40(5):540-51. doi: 10.1080/00365520510012208. PMID 16036506